CLINICAL TRIAL: NCT06786819
Title: Estudo Randomizado de Cluster Escalonado Para Avaliar o Impacto de Uma Plataforma tecnológica Baseada no ERAS (Enhanced Recovery After Surgery) no Tempo de permanência após Cirurgia de revascularização miocárdica: Projeto Tempos Certos - REPLICCAR III
Brief Title: Impact of a Technology Platform Based on Enhanced Recovery After(ERAS) Surgery on Length of Stay After Coronary Artery Bypass Grafting: Timely Project
Acronym: REPLICCARIII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other); Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Instituto do Coração da Universidade de São Paulo, Brazil (Unknown); Hospital Beneficence Portuguese of São Paulo (Unknown); Irmandade Santa Casa Misericórdia Marília (Other); Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Omar Asdrúbal Vilca Mejia, Study Principal Investigator, Head of Quality Improvement in Cardiac Surgery, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5811/24/022
Record Dates: First submitted 2024-11-07; First posted 2025-01-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: ERAS; Cardiac Surgery; Cardiac Surgery-CABG; Digital Health
Keywords: Cardiac Surgery; CABG; ERASCS; ERAS; Digital Health

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care for CABG (No Intervention): Patients will be treated with CABG following the standard of care for each participant institution.
- ERACS with Digital Platform (Experimental): Patient will be treated by the participant institution following a modified protocol based in the ERACS with the aid of a digital platform.
  Interventions: Other: ERACS with Digital Platform

INTERVENTIONS:
Other: ERACS with Digital Platform — The assistance provided to patients in the intervention group will be sequential and prospective. The project will utilize an app based on protocols that prepare patients for rapid recovery (ERAS), starting before surgery and extending up to 30 days post-discharge. This includes pre-operative evaluations (dental, psychological, nutritional, and others), scheduling and confirming hospital admission, and following specific protocols during surgery and intensive care. The app aims to enhance communication and teamwork, improving patient-centered care. It will feature modules for patient and family education, team communication, and activity management through a dashboard. Additionally, it will facilitate interaction with patients through messages and surveys, monitor multidisciplinary team communication, and collect patient-reported outcomes 30 days after the surgical procedure.
  Other Names: ERACS; Enhanced Recovery After Cardiac Surgery; Digital ERAS
  Arms: ERACS with Digital Platform

SUMMARY:
Cardiovascular diseases continue to be the leading cause of death worldwide. Among them, coronary artery disease has the greatest impact, being characterized as one of the main causes of death in Brazil over the last decade. One of the well-established treatments is coronary artery bypass grafting, which is the most performed among cardiac surgeries and, in our scenario, is primarily funded by the Unified Health System (SUS). The information obtained from the Paulista Registry of Cardiovascular Surgeries (REPLICCAR), in partnership with FAPESP, has been important for implementing improvements in the landscape of cardiac surgeries in the state of São Paulo. Although outcomes in cardiac surgery have improved due to the structuring and organization of quality programs, this is still not a reality at the national level. In a situation where data collection and quality initiatives play a central role in continuous improvement, generating value becomes essential for the sustainability of cardiac surgery programs. In this sense, the concept of Enhanced Recovery After Surgery (ERAS) has gained increasing traction. This concept is based on multidisciplinary protocols and scientific evidence, which help prepare patients for rapid recovery, resulting in reduced complications, shorter hospital stays, and, primarily, lower hospital costs. On the other hand, the increase in surgical waiting lists has also led to a rise in home mortality due to cardiac causes. Thus, among the various challenges imposed by the current scenario, the investigators believe that preparing patients for rapid recovery after coronary artery bypass grafting presents an opportunity for the sustainability of the healthcare system. Therefore, the aim of this project is to evaluate the impact of a technology platform based on ERAS on the postoperative recovery time of patients undergoing coronary artery bypass grafting in reference centers in the state of São Paulo, Timely Project - REPLICCAR III.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Indication for primary isolated CABG (elective or urgent status)
* Own a personal cell phone
* Have internet access
* Knowledgeable in using the device
* Full understanding and agreement regarding the informed consent form (ICF)

Exclusion Criteria:

* Indication for associated surgery
* Glycosylated hemoglobin level greater than 8%
* Creatinine clearance less than 30 mL/min
* Pre-operative atrial fibrillation or use of pre-operative anticoagulation
* Hemoglobin less than 12 g/dL
* Users of illicit drugs
* STS score greater than 4%
* Physical or mental disabilities that prevent adherence to the protocol
* Refusal by the patient or family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Lenght of Stay | up to 30 days after surgery
  Compare the length of stay after coronary artery bypass grafting (CABG) with versus without the use of a technology platform based on ERAS.

SECONDARY OUTCOMES:
Percentage of Completeness of Protocol Steps | up to 01 week after surgery.
  Compare adherence to protocol metrics through measure of the execution of the protocol steps by each participant center, during the intervention period. up to one week after surgery.
Morbility and Mortality | up to 6 months after surgery
  Compare morbidity and mortality rates and hospital readmission between the control and intervention groups up to 6 months after CABG.
Patient-reported outcomes (PROM) | up to 6 months after surgery
  Evaluate and patient-reported outcome measures following the questionnaire published by Ben-Ali W, Lamarche Y, Carrier M, Demers P, Bouchard D, El-Hamamsy I, et al. Use of Mobile-Based Application for Collection of Patient-Reported Outcomes in Cardiac Surgery. Innovations: Technology and Techniques in Cardiothoracic and Vascular Surgery. 2021 Nov 1;16(6):536-44. at 01 month and 6 months after surgery.
  This questionary assess self reported pain, quality of recovery, anxiety and engagement of the patient with his/her recovery.
Patient reported experience measure(PREM) | up to 6 months after surgery
  Assessment of patient experience using the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey.

CONTACTS AND LOCATIONS:
Overall Officials: Omar A V Mejia, MD, PhD, Principal Investigator — InCor - Instituto do Coração do Hospital das Clínicas da FMUSP
Locations (1):
- InCor - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borgomoni GB, Reis PH, Pinheiro G, Ribas FF, Silva GSD, Campagnucci VP, Issa M, Farsky PS, Barg MM, Tiveron MG, Dos Reis Falcao LF, Dias RD, Ferreira Lisboa LA, Jatene FB, Mejia OAV. The technological proposal based on enhanced recovery after cardiac surgery for changing traditional care in Latin America: REPLICCAR III Study Protocol. PLoS One. 2025 Dec 31;20(12):e0338301. doi: 10.1371/journal.pone.0338301. eCollection 2025. PMID 41474739